CLINICAL TRIAL: NCT03856255
Title: A Pilot, Single-centered, Single-arm, Feasibility Study Evaluating a Polyp Measurement Device in Patients Undergoing Screening or Surveillance Colonoscopy
Brief Title: Polyp Measurement Device
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19 restrictions with screening/surveillance colonoscopies
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 18-02047
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Results first posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Micro-Tech Endoscopic Gauge (Experimental): Use of the device during screening or surveillance colonoscopy
  Interventions: Device: Micro-Tech Endoscopic Gauge

INTERVENTIONS:
Device: Micro-Tech Endoscopic Gauge — Use of Micro-Tech Endoscopic Gauge to measure any polyp detected during a screening or surveillance colonoscopy.

SUMMARY:
Colorectal cancer is the second-leading cause of cancer death in the United States. Colorectal cancer screening is recommended to begin at age 50 years for most men and women at average risk for this disease. Colonoscopy is a gold standard method of screening for colorectal cancer, allowing for the detection and removal of colorectal polyps, some of which can progress into malignancy. The literature has shown that the removal of polyps during a colonoscopy results in decreased incidence and mortality related to colorectal cancer. Indeed, the last decade has shown a decline in colorectal cancer incidence and mortality in adults over age 50, largely due to increased colonoscopy screening. Currently, the risk of a patient developing colorectal cancer and thus time intervals for colonoscopy surveillance post-polypectomy is determined by the number, pathology, and size of the polyps that are observed and removed during the colonoscopy procedure. Current surveillance guidelines indicate the need for a shorter interval before the next colonoscopy for patients who have one or more polyps that are 10mm or larger. In addition, different polypectomy techniques are indicated for the treatment of polyps less than 20mm in size. For example, cold forceps may be appropriate for removal of 1mm to 2mm polyps, cold snare for polyps less than 10mm, and hot-snare resection for polyps 10mm to 19mm. Yet, while the number and pathology of polyps are easily obtained and verified, it is standard practice for the size of a polyp to be assessed through endoscopist optical visualization alone, without use of an objective device or standard by which to measure it. Often, the endoscopist will compare the size of the polyp to the size of the snare loop to estimate and document the size of the polyp(s). However, with the size of a polyp being a major indicator of malignant potential as well as an indicator of appropriate polypectomy technique and surveillance intervals, a device with which to take and document accurate and objective measurements of polyps during colonoscopy holds the potential for health benefits. In addition to having a potential clinical benefit for each patient in terms of polypectomy and surveillance intervals, as an objective indicator of polyp size, this technique also holds promise for use in future studies that evaluate polyp size as an indicator of potential malignancy (or future malignancy) and for use by national clinical guidelines committees who may utilize these objective data to update future screening and surveillance recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Individuals age 50-85 years old, who require an outpatient screening or surveillance colonoscopy
* Ability to give consent

Exclusion Criteria:

* Pregnancy
* Inflammatory bowel disease

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pochapin, MD, Principal Investigator — New York School of Medicine
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification will be shared. Requests will be directed to mark.pochapin@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol
Time Frame: Data will become available beginning 3 months and ending 5 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal will have access to the data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Micro-Tech Endoscopic Gauge
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Micro-Tech Endoscopic Gauge
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: years] | 63 [50 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 18
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Indicated Ease of Use in Advancing in Measuring Device Catheter Through the Working Channel
Description: Scale of 1-10, with 1 being the easiest and 10 being the hardest
Time Frame: At the time of the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Micro-Tech Endoscopic Gauge
Number analyzed (Participants) | 23
Participants | 21

2. Primary Outcome: Mean Score Indicating Ease of Extending and Retracting the Device
Description: Scale of 1-10, with 1 being the easiest and 10 being the hardest
Time Frame: At the time of of the procedure
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Micro-Tech Endoscopic Gauge
Number analyzed (Participants) | 23
score on a scale | 1.43 (0.21)

3. Primary Outcome: Mean Score Indicating Ease of Use in Placing the Measuring Device Adjacent to the Polyp in Order to Determine a Measurement
Description: Scale of 1-10, with 1 being the easiest and 10 being the hardest
Time Frame: At the time of the procedure
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Micro-Tech Endoscopic Gauge
Number analyzed (Participants) | 23
score on a scale | 2.62 (0.40)

4. Primary Outcome: Mean Score Indicating Ease of Use in Taking a Picture That Included the Measuring Device and Polyp in Order to Photo-document the Measurement Reading
Description: Scale of 1-10, with 1 being the easiest and 10 being the hardest
Time Frame: At the time of the procedure
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Micro-Tech Endoscopic Gauge
Number analyzed (Participants) | 23
score on a scale | 2.17 (0.87)

5. Secondary Outcome: Mean Difference in Size of Polyp
Description: The size of the polyp measured by the device will be subtracted from the size of the polyp as measured by the standard, device-free optical visualization.
Time Frame: At the time of the procedure
Measure: Mean (Standard Error); unit: mm
Arm/Group | Micro-Tech Endoscopic Gauge
Number analyzed (Participants) | 23
mm | 0.28 (0.21)

ADVERSE EVENTS:
Time Frame: 24 hours after procedure
Arm/Group | Micro-Tech Endoscopic Gauge
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT03856255/Prot_SAP_000.pdf